CLINICAL TRIAL: NCT02913092
Title: Electronic Monitoring of Medication Adherence in Moderate to Severe Asthma
Brief Title: Electronic Monitoring of Medication Adherence in Moderate to Severe Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Stony Wold-Herbert Fund, Inc. (Other)
Responsible Party: Principal Investigator, Marina Reznik, Associate Professor of Pediatrics, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016-7001; Community Service Award (Other Grant/Funding Number: Stony Wold-Herbert Fund)
Record Dates: First submitted 2016-09-18; First posted 2016-09-23 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic sensor and OW education (Experimental): MDI sensor-generated alerts will be relayed and responded to (e.g. outreach worker contacts the participant for a missed dose) in real-time to the intervention group. Outreach worker will also assess intervention group participants' need for further asthma education and provide asthma education over the phone
  Interventions: Behavioral: Electronic sensor and OW education
- Usual Care (No Intervention): Usual care group will receive the electronic tracker but the sensor-generated alerts will not be delivered. If the usual care group rescue inhaler data reveals frequent use of rescue medication (daily use for >3 days) investigators will reach out (via app or phone call) to advise the participant to see their physician

INTERVENTIONS:
Behavioral: Electronic sensor and OW education — MDI sensor-generated alerts will be relayed via app platform on participant's phone and responded to (e.g. outreach worker contacts the patient for a missed dose) in real-time to the intervention group. Outreach worker will also assess intervention group participants' need for further asthma education and provide education over the phone
  Arms: Electronic sensor and OW education

SUMMARY:
This study will evaluate the role of using electronic sensors for asthma inhaler devices in monitoring medication adherence and asthma control

DETAILED DESCRIPTION:
This study will assess the feasibility of using electronic sensors for asthma inhalers in a population of urban minority adults and children with moderate-severe asthma in the Bronx.

Investigators will also assess differences in asthma outcomes (specifically asthma control as a primary outcome measure) and treatment adherence in a group of participants with moderate-severe asthma who use inhalers with electronic sensors and real-time remote outreach worker monitoring/feedback compared to a group of participants who use inhalers with electronic sensors but without real-time monitoring/feedback.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) and children (5-11 years old) with a clinical history (i.e. physician-diagnosed) of asthma
* Moderate to severe asthmatics with ≥1 asthma-related ED visits or hospitalizations in the past year
* Use of daily controller inhaler medications
* Adult non-smokers, or lifetime use <5 pack years with no smoking in last 1 yr
* Smartphone required
* English or Spanish speaking

Exclusion Criteria:

* No smartphone
* Use of oral corticosteroids in prior 4 weeks
* Pregnancy
* Psychiatric conditions

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test | change from baseline to 6 months
  validated asthma control measure

SECONDARY OUTCOMES:
Medication adherence | change from baseline to 6 months
  measured by electronic sensor
Health care utilization | change from baseline to 6 months
  ED visits and hospitalizations will be assessed via electronic health records

CONTACTS AND LOCATIONS:
Overall Officials: Marina Reznik, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No